CLINICAL TRIAL: NCT05031026
Title: Dexmedetomidine Infusion to Prevent Hepatic Ischemia-reperfusion Injury-induced Glycocalyx Degradation and Early Allograft Dysfunction in the Sitting of Adult Living Donor Liver Transplantation
Brief Title: Dexmedetomidine to Prevent Hepatic Ischemia-reperfusion Injury-induced Glycocalyx Degradation and Early Allograft Dysfunction in Liver Transplantation
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aboubakr Youssef Ahmed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AYA1
Record Dates: First submitted 2021-08-17; First posted 2021-09-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplant; Complications
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- donor group (Active Comparator): where donors only will receive dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- recpient group (Active Comparator): where recepients only will receive dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- control group (Placebo Comparator): both donors and recipients will receive a placebo
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine infusion rule in prevention of IRI
  Other Names: Precedex
  Arms: donor group; recpient group
Drug: Normal Saline — normal saline infusion as a placebo
  Other Names: NS 0.9%
  Arms: control group

SUMMARY:
the aim of the study is to approve the hypothesis that dexmedetomidine can protect against glycocalyx degradation induced by hepatic ischemia-reperfusion injury and hence can reduce the subsequent complications as early allograft dysfunction, other organ dysfunction and hemodynamic instability

DETAILED DESCRIPTION:
The endothelial glycocalyx (EGCX) is a carbohydrate conjugate. It forms the vascular endothelial surface layer and is an important mediator of vascular permeability, coagulation, and inflammation. Inflammation, ischemia reperfusion, diabetes, and hypervolemia can cause EGCX damage.

When the EGCX is damaged by different mechanisms, glycocalyx-shedding products can be measured in the plasma. Syndecan-1 and heparan sulfate are two of components of the endothelial glycocalyx that have increased plasma concentrations after glycocalyx injury. The amount of glycocalyx-shedding correlates with the severity of the underlying pathological condition as different studies have shown.

The EGCX is an important target in the pathophysiological process of ischemia-reperfusin injury (IRI). Its destruction appears to play a central pathophysiological role in the development of IRI in conditions like shock, myocardial infarction, stroke, traumatic blood loss and during solid organ transplantation.

That damage to the endothelial glycocalyx significantly contributes to the development of IRI as recent studies have suggested. Schiefer et al. reported significantly higher plasma levels of syndecan-1 in liver graft recipients after transplantation than before transplantation, indicating destruction of the endothelial glycocalyx.

In animal studies, various drugs that may protect and/or restore the endothelial glycocalyx have been tested, while human trials are still lacking. Glycocalyx-protective strategies have been investigated during major surgery and the results indicated that preventive measures may be effective against glycocalyx destruction.

Dexmedetomidine is a potent and highly selective α2 adrenoreceptor agonist. It is widely used for sedation in ICU and also offers a good perioperative hemodynamic stability and an intraoperative anesthetic- sparing effect. So, it is used as an anesthetic adjuvant during surgery. Some studies have applied it for postoperative sedation in the setting of liver transplantation. Experimentally, it has a favorable effect on liver tissues in case of sepsis. It is also reported to have protective effects against IRI of the heart, kidney, brain, testis and recently against IRI of the liver.

The protective effects of dexmedetomidine against liver injury induced by ischemia and reperfusion during adult Liver transplantation, are indicated by suppression of the serum Intercellular adhesion molecule-1 (ICAM-1) levels, better scores of histopathological assessment, and augmented postoperative liver function tests.

The activation of α2 adrenoreceptors might be attributable to anti-inflammatory, anti-oxidant, and other cellular protective properties.

The protection might be also attributable to the enhancement of Nuclear factor, erythroid 2 like 2 (Nrf2) pathway and the suppression of mitogen-activated protein kinase (MAPK), Caspase-3/Poly (ADP-Ribose) polymerase (PARP), and Toll-like receptor 4 (TLR4)/NF-κB pathways.

In the clinical setting, a randomized controlled trial by Wang et al. of 44 patients undergoing hepatectomy found that intraoperative treatment with dexmedetomidine resulted in lower serum ALT and AST levels in the first 72 hours postoperatively.

Another study conducted in rats found that dexmedetomidine inhibited the decrease of EGCX thickness and the increase of the blood level of syndecan-1 which induced by heat stroke, which suggests that dexmedetomidine may have a protective action for EGCX.

To the investigators knowledge and till 2021, no previous human studies had discussed the protective effect of dexmedetomidine against glycocalyx degradation induced by hepatic ischemia-reperfusion injury and its impact on early allograft dysfunction in the sitting of adult living donor liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-60 years.
2. Model for end-stage liver disease (MELD) score 12-20.
3. No severe hemodynamic instability.
4. The liver donors aged 18-50 years and the sum of macro- and microvesicular hepatic steatosis has to be less than 30%.

Exclusion Criteria:

1. History of psychiatric/neurological illness.
2. Cardiovascular disease.
3. Hypertensive patients.
4. Morbid obese patients (body mass index (BMI) > 35).
5. Chronic obstructive pulmonary disease; pulmonary dysfunction (PaO2 less than 60 mmHg).
6. Known allergic reaction to any of the study medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
syndecan-1 level | 48 hours
  Change in syndecan-1 level 5 minutes after hepatic artery declamping

SECONDARY OUTCOMES:
Incidence of Primary nonunction (PNF) which is defined as graft loss, retransplantation, or participant death due to graft non-function in first 30 days without detectable technical or immunological problems. | 30 days
  Number of patients developed PNF
Incidence of acute kidney injury ( AKI ) during postoperative days 1-7. | 7 days
  Number of patients developed AKI: AKI is defined as a rise in creatinine of ≥50% from its baseline value and/or a fall in the glomerular filtration rate (GFR) by ≥25%, and/or a decrease in urine output below 0.5 ml/kg/h for 6 h or more
Incidence of acute respiratory distress syndrome ( ARDS ) during postoperative days 1-7. Defined according to Berlin modification of the American European Consensus Committee (AECC) definitions published in 2012 | 7 days
  Number of patients developed ARDS
duration of post-operative mechanical ventilation | 30 days
  Time on MV
ICU and hospital stay after surgery. | 60 days
  Time in hospital
All-cause 30-day mortality | 30 days
  Mortality occurance
Incidence of early hepatic allograft dysfunction ( EAD ) Defined according to Olthoff's criteria published in 2010: (1) bilirubin ≥10 mg/dL on day 7, or (2) INR > 1.6 on day 7, or (3) AST/ ALT > 2000 IU/L within first 7 days | 7 days
  Number of patients developed allograft dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Zhu YX, Zhou JH, Li GW, Zhou WY, Ou SS, Xiao XY. Dexmedetomidine protects liver cell line L-02 from oxygen-glucose deprivation-induced injury by down-regulation of microRNA-711. Eur Rev Med Pharmacol Sci. 2018 Oct;22(19):6507-6516. doi: 10.26355/eurrev_201810_16065. PMID 30338821
- [Background] Nieuwdorp M, van Haeften TW, Gouverneur MC, Mooij HL, van Lieshout MH, Levi M, Meijers JC, Holleman F, Hoekstra JB, Vink H, Kastelein JJ, Stroes ES. Loss of endothelial glycocalyx during acute hyperglycemia coincides with endothelial dysfunction and coagulation activation in vivo. Diabetes. 2006 Feb;55(2):480-6. doi: 10.2337/diabetes.55.02.06.db05-1103. PMID 16443784
- [Result] Mathis S, Putzer G, Schneeberger S, Martini J. The Endothelial Glycocalyx and Organ Preservation-From Physiology to Possible Clinical Implications for Solid Organ Transplantation. Int J Mol Sci. 2021 Apr 13;22(8):4019. doi: 10.3390/ijms22084019. PMID 33924713
- [Result] Fayed NA, Sayed EI, Saleh SM, Ehsan NA, Elfert AY. Effect of dexmedetomidine on hepatic ischemia-reperfusion injury in the setting of adult living donor liver transplantation. Clin Transplant. 2016 Apr;30(4):470-82. doi: 10.1111/ctr.12713. Epub 2016 Mar 3. PMID 26856320